CLINICAL TRIAL: NCT04759092
Title: A Four Month Home Based tDCS Study on Patients With Alzheimer's Disease.
Acronym: tDCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: University of Tromso (Other)
Responsible Party: Principal Investigator, Ole Kristian Grønli, MD/phd senior consultant, University Hospital of North Norway
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TDCS1HB
Record Dates: First submitted 2021-01-28; First posted 2021-02-18 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Treatment study, open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with tDCS (Experimental): Home based treatment with tDCS for four months
  Interventions: Device: transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: transcranial direct current stimulation (tDCS) — Apply 30min low dose (2mA) transcranial current stimulation on the scalp every day for four months.
  Other Names: tDCS

SUMMARY:
The study is an open label study on patients with Alzheimer's dementia using home based transcranial direct current (tDCS) stimulation. Aims of the study is to investigate applicability and effect of treatment.

DETAILED DESCRIPTION:
Active tDCS of 2mA is applied via surface based electrodes daily for 30 minutes over a 4 month period. Anodal electrode is placed over the left temporal lobe. Participants is followed up by home visit and phone calls.

Cognitive tests are performed prior to the treatment period, right after finishing 4 months of treatment and 4 months after treatment is terminated.

ELIGIBILITY:
Inclusion Criteria:

* Age 60-85.
* Fulfil diagnostic criteria of probable Alzheimer's dementia.
* Participants has to live with a caregiver.
* If medicated with cholinesterase inhibitors or memantine, a stable dose the last three months before inclusion is required.

Exclusion Criteria:

* Implant in head
* Seizure history
* Severe illness,
* Psychosis or depression measured with a cornell score over 11.
* Mini mental status (MMSE) score<17.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
To investigate adverse effects of the treatment | 4 months
  Investigation of tolerability of long term home based tDCS to patients with Alzheimer's by using the Adverse effect questionnaire for tDCS
To investigate effect of the treatment | 8 months
  Investigate possible change in cognitive tests (Repeatable Battery for the Assessment of Neuropsychological Status (RBANS), Mini Mental Status Examination ( MMSE), Clock drawing test, Trail making test A & B) after 4 months treatment and change 4 months after end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ole K Grønli Grønli, MD/PHD, Principal Investigator — University Hospital of North Norway
Locations (1):
- University Hospital of North Norway, Tromsø, Troms, Norway

IPD SHARING:
Plan to Share IPD: No
No plan of sharing individual participant data, because its not a part of the approvement of the advisory board.

REFERENCES:
- [Derived] Gronli OK, Daae Rasmussen I, Aslaksen PM, Bystad M. A four-month home-based tDCS study on patients with Alzheimer's disease. Neurocase. 2022 Jun;28(3):276-282. doi: 10.1080/13554794.2022.2100710. Epub 2022 Jul 19. PMID 35852094